CLINICAL TRIAL: NCT05644600
Title: An Open Label, Randomised Study in Healthy Participants to Investigate the Effect of AZD5055 on the Pharmacokinetics of Nintedanib.
Brief Title: A Study to Assess the Effect of AZD5055 on the Pharmacokinetics (PK) of Nintedanib in Healthy Participants.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated as no drug-drug interactions were observed in Part-A of the study and therefore Part-B of the study was not required as per protocol.
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D8960C00003; 2022-003116-84 (EudraCT Number)
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Healthy Subjects
Keywords: Drug-drug interaction; Idiopathic pulmonary fibrosis; Interstitial lung diseases with progressive fibrosis; Porcupine inhibitor; Pharmacokinetics
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — nintedanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment A (Experimental): The subjects will receive Nintedanib soft capsules, fasted state.
  Interventions: Drug: Nintedanib
- Treatment B (Experimental): The subjects will receive dose B of the oral suspension of AZD5055 immediately followed by nintedanib in the fasted state.
  Interventions: Drug: Nintedanib; Drug: AZD5055
- Treatment C (Experimental): The subjects will receive dose C of the oral suspension of AZD5055 immediately followed by nintedanib in the fasted state.
  Interventions: Drug: Nintedanib; Drug: AZD5055
- Treatment D (Experimental): The subjects will receive dose C of the oral suspension of AZD5055 4 hours after nintedanib in the fasted state.
  Participants would remain in the fasted state until 1.5 hours after AZD5055 administration.
  Interventions: Drug: AZD5055

INTERVENTIONS:
Drug: Nintedanib — The subjects will be administered Nintedanib soft capsules single oral dose in the morning of Day 1 in fasted state.
  Arms: Treatment A; Treatment B; Treatment C
Drug: AZD5055 — The subjects will be administered AZD5055 as single oral dose on Day 1 in the fasted state.
  Arms: Treatment B; Treatment C; Treatment D

SUMMARY:
The study is intended to quantify the effect of co-administration and staggered dosing of AZD5055 and nintedanib on exposures of nintedanib in healthy participants.

DETAILED DESCRIPTION:
This study will be an open-label, randomised, crossover study in healthy participants (males and females of non-childbearing potential).

The study will comprise two parts: Part A and Part B.

The study will include a screening period of 28 days for both Part A and Part B.

Part A will be a 3-period (Periods 1, 2, 3), 3-treatment (Treatments A, B, C) crossover study, performed at a single clinical unit. During the 3 periods (Periods 1, 2, 3) participants will participate from Day -1 of Period 1 to 72 hours after the nintedanib dose in Period 3. In each period, the participants will receive AZD5055 immediately before the nintedanib dose in the morning of the first day. In Part A, all participants will be randomised to one of 3 sequences.

An interim analysis of data from Part A will be performed, and Part B (conducted only if an interaction between AZD5055 and nintedanib is observed in Part A) will be a 2-period (Periods 1, 2), 2-treatment (Treatments A, D) crossover study, performed at 2 clinical units. In each period, the participants in Treatment D will be dosed with AZD5055 4 hours after the nintedanib dose in the morning of the first day. In Part B, all participants will be randomised to one of 2 sequences.

For both Part A and Part B, there will be a minimum washout period of approximately 72 hours between each AZD5055 dose administration. And, a follow-up visit will be performed, at 6 ± 1 days after the last dose of nintedanib in last period.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy nonsmoking male and female (of non-childbearing potential) participants aged 18 to 55 years (inclusive) with suitable veins for cannulation or repeated venipuncture.
2. Females must have a negative pregnancy test, must not be lactating and must be of non childbearing potential.
3. Male participants and their woman partners of childbearing potential must be willing to use highly effective contraception measures and must refrain from donating sperm or fathering a child.

Exclusion Criteria:

1. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the study, or influence the results or the participant's ability to participate in the study.
2. History or presence of chronic gastrointestinal, hepatic, or renal disease, any acute disease in these organs, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
3. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of IMP (Investigational Medicinal Product).
4. Untreated TB (Tuberculosis) or a positive result for the IGRA (Interferon Gamma Release Assay) (ie, QuantiFERON TB Gold).
5. Individuals with chronic infections (eg, urinary tract infection) or who are at increased risk of infection (eg, surgery, trauma, severe dental disease, or significant infection) .
6. History of severe COVID-19 (corona virus) infection requiring hospitalisation within the last 12 months prior to Screening, or clinical history compatible with Long COVID-19 (symptoms beyond 12 weeks of acute infection).
7. Has received live or live attenuated vaccine in the 30 days prior to dosing, the first dose of COVID-19 vaccine within 30 days prior to randomisation, or a COVID-19 vaccine second or booster vaccination within 10 days of Screening.
8. History of osteoporosis, osteomalacia, Paget's disease of the bone, thyrotoxicosis, rheumatoid arthritis, Cushing's disease, or a pathological fracture.
9. History of a traumatic fracture within 6 months of Screening.
10. Any laboratory values with the following deviations:

(1) Alanine aminotransferase > ULN (2) Aspartate aminotransferase > ULN (3) Total bilirubin > ULN (4) White blood cell count < 3.5 × 109/L (5) Platelet < LLN (6) eGFR < 90 ml/min/1.73 m2 (Cockroft-Gault or CKD-EPI formula) 11. Any clinically important abnormalities in rhythm, conduction, or morphology of the resting ECG (Electrocardiogram) and any clinically important abnormalities in the 12-lead ECG .

12. Any positive result on Screening for active hepatitis A, hepatitis B surface antigen, hepatitis B core antibody, hepatitis C antibody, or HIV antibody, or any known chronic/active liver diseases.

13. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD5055 or nintedanib.

14. Use of any prescribed or non prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of IMP or longer if the medication has a long half life.

15. Subjects who have previously received AZD5055.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2023-05-26 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2023-07-17 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma (peak) drug concentration (Cmax) | Day 1 - 9
  The effect of AZD5055 on the PK of nintedanib alone and in combination AZD5055 will be assessed.
Area under plasma concentration time curve from zero to infinity (AUCinf) | Day 1 - 9
  The effect of AZD5055 on the PK of nintedanib alone and in combination AZD5055 will be assessed.
Area under the plasma concentration time curve from zero to the last quantifiable concentration (AUClast) | Day 1 - 9
  The effect of AZD5055 on the PK of nintedanib alone and in combination AZD5055 will be assessed.

SECONDARY OUTCOMES:
Cmax of AZD5055 (Part A only) | Day 1-9
  The PK of AZD5055 after single Dose B or Dose C doses administered with a single oral dose of nintedanib will be evaluated.
AUCinf of AZD5055 (Part A only) | Day 1-9
  The PK of AZD5055 after single Dose B or Dose C doses administered with a single oral dose of nintedanib will be evaluated.
AUClast of AZD5055 (Part A only) | Day 1-9
  The PK of AZD5055 after single Dose B or Dose C doses administered with a single oral dose of nintedanib will be evaluated.
Cmax of ninetedanib alone and in combination AZD5055 (Part B only) | Day 1-6
  The effect of AZD5055 on the PK of nintedanib when AZD5055 dose is staggered (delayed) 4 hours is assessed.
AUCinf of ninetedanib alone and in combination AZD5055 (Part B only) | Day 1-6
  The effect of AZD5055 on the PK of nintedanib when AZD5055 dose is staggered (delayed) 4 hours is assessed.
AUClast of ninetedanib alone and in combination AZD5055 (Part B only) | Day 1-6
  The effect of AZD5055 on the PK of nintedanib when AZD5055 dose is staggered (delayed) 4 hours is assessed.
Number of subject with Adverse event (AE) and serious Adverse event (SAE) | SAEs: From Screening (Day -28 to -2) to Day -1 of Period 1 AEs: From Day 1 untill follow up (Day 13)
  The safety and tolerability following single oral doses ofAZD5055 administered with nintedanib in healthy participants will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Glendale, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual subject-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual subject-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home